CLINICAL TRIAL: NCT03097003
Title: An Observational Study of the Real-life Management of Psoriasis Patients Treated With Otezla® (Apremilast) in Belgium
Brief Title: A Study of the Real-life Management of Psoriasis Patients Treated With Otezla® (Apremilast) in Belgium
Acronym: OTELO
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-10004-PSOR-016; U1111-1194-1580 (Other: WHO)
Record Dates: First submitted 2017-03-24; First posted 2017-03-31 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Psoriasis
Keywords: Proriasis; Real-life management; Observational; Otezla; CC-10004; Apremilast; Belgium; OTELO
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Use of Apremilast in patient with plaque psoriasis: Psoriasis patients treated with Otezla® (Apremilast) in Belgium
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Psoriasis patients treated with Otezla® (Apremilast) in Belgium

SUMMARY:
OTELO is a national (Belgium), multicentre, prospective, non-interventional, post-marketing study. The study will include a representative sample of approximately 250 patients with moderate-to-severe plaque psoriasis for whom the treating dermatologist has decided to begin apremilast treatment in accordance with the local label and reimbursement criteria. Patients may be enrolled into the study up to 4 weeks after commencing the study treatment.

As this study is non-interventional, drug dosing and treatment duration will be at the sole discretion of the treating dermatologist, in accordance with the local label and daily clinical practice.

DETAILED DESCRIPTION:
Patient care will follow routine clinical practice, involving regular follow-up visits, without any mandatory visit. In daily practice, patients are usually seen by their treating dermatologists every 3 months. In this study, patients will be followed-up for a least 6 months and at most 18 months after apremilast treatment initiation. Patient data will be collected until 31st December 2018. Assuming a recruitment phase of 18-month duration starting as of December 2016, individual patient follow-up times will range from 6 to 18 months, depending on the inclusion date. During the first months of the study, the recruitment rate has been slower than expected. Therefore, it has been decided in October 2017 to increase the period of recruitment to 18 months in order to have enough evaluable patients to keep the accuracy required for the statistical analysis.

During the study, it is expected to collect data at inclusion and at 6 months after apremilast initiation in all patients. As per NIHDI recommendations, patients should consult their treating dermatologists 6 months after apremilast initiation in order to evaluate treatment response and decide on treatment continuation for an additional period of 12 months. For patients recruited early in the study, data will be collected during the next follow-up visits up to 18 months after apremilast initiation. Only data pertaining to visits occurring at 9 (± 1), 12 (± 1), 15 (±1), and 18 (± 1) months after treatment initiation will be collected. If a study visit occurs approximately 3 (± 1) months after treatment initiation, the data will also be recorded.

All clinical data collected during this non-interventional study will be routinely documented in the patient's medical records, which are the main source of information. The study data will be collecting via an eCRF. Data from source documents including PRO-questionnaires will be entered in the eCRF by the investigator or other authorised appropriately designed and trained study site personnel. Data entered into the eCRF will be reviewed for consistency by the Data Manager using both automated logical checks (issuing in automatic queries generated by the system) and manual review (issuing in manual checks set by the Data Manager or the Monitor into the eCRF). All data collected within the eCRF will be approved and electronically signed and dated by the Investigator or designee. At the conclusion of the study, before the final statistical analysis, the eCRF and other study data will be locked to further additions or corrections.

During the study, the Clinical Research Associate (CRA) will contact each study site on a regular basis in order to check the progress and conduct of the study. If issues regarding study conduct arise, additional on-site visits may be performed. In particular, a quality analysis will also be performed and based on data quality, it will be decided whether on-site monitoring is necessary, for which site and on which percentage of patients. During monitoring visits, eCRFs, patient's source documents, and all other study documentation will be reviewed by the CRA. Accuracy will be checked by performing source data verification that is a direct comparison of the entries made onto the eCRF against the appropriate source documentation.

Adverse events AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) terminology. The detailed methodology of the statistical analyses will be documented in a statistical analysis plan (SAP). The SAP will be written by the Clinical Research Organisation (CRO) in charge of the study and will be validated by sponsor prior to performing the analysis and obligatory before the database lock. A scientific committee has been selected for this study. This committee will provide advice on the SAP.

ELIGIBILITY:
Inclusion Criteria:

- Patients who meet ALL the following criteria can be enrolled:

* Male or female aged at least 18 years.
* With a diagnosis of moderate-to-severe chronic plaque psoriasis. As per Belgian National Institute for Health and Disability Insurance (NIHDI), moderate-to-severe plaque psoriasis in adult patients is defined by a Body Surface Area (BSA) > 10% or aPsoriasis Area and Severity Index (PASI) > 10.
* For whom the treating dermatologist has made the decision to commence apremilast treatment in accordance with the local label and reimbursement criteria
* Able to follow the instructions of the study.
* Having signed an Informed Consent Form (ICF)

Exclusion Criteria:

Patients who meet AT LEAST one of the following exclusion criteria will be excluded:

* Patients who have received apremilast > 4 weeks prior to the enrolment visit.
* Women who are pregnant, breastfeeding or planning on becoming pregnant.
* Non-menopausal women who are not using an adequate contraception method.
* Patients with hypersensitivity to apremilast or to one of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with moderate-to-severe plaque psoriasis visiting dermatology practices in Belgium and eligible for treatment with apremilast according to the local label and reimbursement criteria.
  Patients may be enrolled into the study up to 4 weeks after commencing the treatment with apremilast. The decision to treat the patient with apremilast will be made prior to the decision to enter the patient into the study.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Patient Benefit Index for skin diseases (standard version) (PBI-S) ≥ 1 at 6 months after apremilast initiation. | Up to 6 Months
  The PBI-S questionnaire for skin diseases is a validated instrument to assess treatment needs and benefits in patients with skin diseases. It comprises 23 items on patient-relevant therapy needs and benefits.

SECONDARY OUTCOMES:
Characteristics of the patients treated with apremilast | Baseline
  The patients treated with Apremilast will be described according to the following characteristics: demographics (age, gender, weight, height, and ethnicity), professional status, lifestyle habits, medical history (including psoriasis treatment history), and comorbidities
Proportion of patients with PBI-S = 4 at 6 months after apremilast initiation | Up to 6 Months
  The PBI-S questionnaire for skin diseases is a validated instrument to assess treatment needs and benefits in patients with skin diseases. It comprises 23 items on patient-relevant therapy needs and benefits.
PBI-S outcome score after apremilast initiation | up to 18 months
  The PBI-S questionnaire for skin diseases is a validated instrument to assess treatment needs and benefits in patients with skin diseases. It comprises 23 items on patient-relevant therapy needs and benefits.
Proportion of patients having clear/no psoriasis based on Patient Global Assessment (PtGA) at 6 months after apremilast initiation | up to 6 months
  PtGA is defined as single-item 5-point categorised scale reflecting the patient's overall impression of psoriasis severity. This scale ranges from 0 (clear/no psoriasis) to 4 (severe psoriasis)
Change from baseline in the PtGA after apremilast initiation | up to 18 months
  PtGA is defined as single-item 5-point categorised scale reflecting the patient's overall impression of psoriasis severity. This scale ranges from 0 (clear/no psoriasis) to 4 (severe psoriasis)
Proportion of patients with Dermatology Life Quality Index (DLQI) ≤ 5 at 6 months after apremilast initiation. | Up to 6 Months
  DLQI is 10-item validated questionnaire used in a wide range of dermatological conditions and across a wide range of disease severity as a quality of life instrument. It covers a variety of health dimensions, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Each item is graded on a Likert scale of 0-3, which gives an overall score ranging from 0 to 30 where lower scores mean better quality of life.
Change from baseline in the DLQI score after apremilast initiation | up to 18 months
  DLQI is 10-item validated questionnaire used in a wide range of dermatological conditions and across a wide range of disease severity as a quality of life instrument. It covers a variety of health dimensions, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Each item is graded on a Likert scale of 0-3, which gives an overall score ranging from 0 to 30 where lower scores mean better quality of life.
Change from baseline in the psoriasis symptomatology | up to 18 months
  Psoriasis symptomatology - pruritus, scalp psoriasis, nail psoriasis, skin discomfort/pain, joint pain, fatigue, overall wellbeing. Each symptom will be graded using a 7-grade discrete rating scale
Change from baseline in the patient-reported treatment satisfaction (TSQM-9) | up to 18 months
  TSQM-9 is 9-item validated self-administered questionnaire used to evaluate the patient's overall satisfaction with study treatment. The TSQM-9 consists of 8 items that make up 3 specific scales (effectiveness, side effects, convenience) and one global satisfaction scale. Scale scores are transformed into scores from 0 to 100 with higher scores representing higher satisfaction in that domain.
Proportion of patients achieving Psoriasis Area and Severity Index (PASI) 50 or PASI 75 at 6 months after apremilast initiation | Up to 6 Months
  PASI is common clinical tool used to measure the severity and extent of psoriasis. PASI score is a composite score grading the severity of psoriasis in four body regions according to erythema, scaling, and thickness, and the total area of skin affected. The final composite score ranges from 0 to 72, with a higher score indicating a greater severity of psoriasis. PASI 50 and PASI 75 responses were defined as >=50% and >= 75% improvement in overall PASI score when compared to baseline
Change from baseline in the disease activity scores in terms of Body Surface Area (BSA) | up to 18 months
  BSA is measurement of the body area involved in relation to the whole body surface.
Change from baseline in the disease activity scores in terms of PASI | up to 18 months
  PASI is common clinical tool used to measure the severity and extent of psoriasis. PASI score is a composite score grading the severity of psoriasis in four body regions according to erythema, scaling, and thickness, and the total area of skin affected. The final composite score ranges from 0 to 72, with a higher score indicating a greater severity of psoriasis. PASI 50 and PASI 75 responses were defined as >=50% and >= 75% improvement in overall PASI score when compared to baseline
Mean duration of apremilast treatment in biologic-naïve patients and in patients having received a previous biological treatment | Up to 18 Months
  Time to the stop of the treatment by Apremilast will be calculated as the time interval from the date of apremilast initiation to the date of the apremilast stop
Rate of discontinuation of apremilast treatment within 6 months after initiation | Up to 6 months
  Descriptive statistics will be provided for the rate and reasons for discontinuation of treatment within 6 months. This analysis will be performed on safety population and restricted to patients who stop the treatment before the time point to analyse or for which the follow-up is at least so long as the time point to analyse.
Adverse Events (AEs) | Up to 18 months
  Number of participants with adverse event

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (22):
- Belgium (22):
  - AZ Sint Jan, Bruges
  - CHU St Pierre, Brussels
  - CHU Brugmann (Victor Horta), Brussels
  - Clin Univ de Bxl Hôpital Erasme, Brussels
  - UZ Brussel, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Antwerpen, Edegem
  - Private Practice Geel, Geel
  - Private Practice Genk, Genk
  - AZ Sint Lucas, Ghent
  - UZ Gent, Ghent
  - CHU UCL Mont-Godinne, Godinne
  - Clinique André Renard d'Herstal, Herstal
  - Private Practice Lede, Lede
  - UZ Leuven Sint Rafael, Leuven
  - CHU Sart-Tilman, Liège
  - GHdC - site IMTR, Loverval
  - Dermatologie Maldegem, Malgegem
  - Private Practice Mons, Mons
  - Private Practice Namur, Namur
  - Ste Elisabeth - Namur, Namur
  - CH Bois Abbaye-Hesbaye, Seraing

REFERENCES:
- [Derived] Ghislain PD, Lambert J, Lam Hoai XL, Hillary T, Roquet-Gravy PP, de la Brassinne M, Segaert S. Real-Life Effectiveness of Apremilast for the Treatment of Psoriasis in Belgium: Results From the Observational OTELO Study. Adv Ther. 2022 Feb;39(2):1068-1080. doi: 10.1007/s12325-021-01981-7. Epub 2022 Jan 3. PMID 34977985
- See also: Expanded Access for CC-10004 — https://clinicaltrials.gov/ct2/show/NCT03097003?term=CC-10004-PSOR-016&rank=1